CLINICAL TRIAL: NCT07279168
Title: Investigation of the Effectiveness of Virtual Reality (VR) Hypnosis in Improving Poor Sleep Among Chinese Childhood Cancer Survivors: A Mixed Methods Randomized Controlled Trial
Brief Title: Investigation of the Effectiveness of Virtual Reality (VR) Hypnosis in Improving Poor Sleep Among Chinese Childhood Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Research Grants Council, Hong Kong (Other); Hong Kong Children's Hospital (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Virtual reality (VR) hypnosis
Record Dates: First submitted 2025-11-19; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Cancer
Keywords: virtual reality hypnosis; Chinese childhood cancer survivors; sleep
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT-I (Active Comparator)
  Interventions: Behavioral: CBT-I
- VR relaxation (Other): The same length and delivery mode as VR hypnosis, but without a hypnosis component. The VR relaxation group will allow us to distinguish the effects of VR from those of VR hypnosis.
  Interventions: Behavioral: VR relaxation
- VR hypnosis (Experimental)
  Interventions: Behavioral: VR hypnosis

INTERVENTIONS:
Behavioral: VR hypnosis — Participants will individually complete VR hypnosis, comprising six 30-minute sessions, conducted by a clinical psychologist on 6 consecutive Saturdays in Hong Kong Children's Hospital or home depend on participants' preference. Participants will be asked to wear head-mounted glasses which can display different scenarios. The participant will select one scenario on the basis of preference. In phase 1 (induction), a narrator will ask the participant to complete various tasks, such as naming animals that participants see. In phase 2 (deepening), the glasses will continue to show the relaxing scenery, with the narrator guiding the participant to pay attention to their breathing and muscle movements. In phase 3 (suggestion), participants will be guided to change negative thoughts and behaviors arising in response to poor sleep. In phase 4 (reawakening), the participants will be guided to return to the peaceful scene with a renewed sense of focus, such that participants will sleep well.
  Arms: VR hypnosis
Behavioral: VR relaxation — Participants will take part in a VR relaxation intervention supervised by a research assistant in Hong Kong Children's Hospital or participants' home depend on participants' preference, which comprises six 30-minute sessions, will be conducted on 6 consecutive Saturdays. The head-mounted display will show five relaxing scenarios (exploring an island, walking through a forest, observing different animals, climbing a mountain, and swimming in the sea), but without a hypnosis component.
  Arms: VR relaxation
Behavioral: CBT-I — It will have six 30-minute sessions delivered by a clinical psychologist in Hong Kong Children's Hospital or home depend on participants' preference on six consecutive Saturdays in a standard sequence: (1) psychoeducation which provides information on sleep, its function and characteristics, (2) sleep hygiene, in which guidelines that promote healthy sleep are followed, (3) stimulus control, which breaks the association between bedtime and anxiety by avoiding any activities in bed not related to sleep; (4) sleep restriction, which limits the amount of time in bed to increase the sleep drive, and (5) cognitive restructuring, which replaces negative thoughts of sleep with constructive thoughts; and (6) relaxation techniques that can quiet the mind and the body in preparation for sleep. A sleep diary will be provided along with handouts and worksheets for skill acquisition and practice.
  Arms: CBT-I

SUMMARY:
The study aims to examine the effectiveness of virtual reality (VR) hypnosis for improving sleep in among Chinese childhood cancer survivors. Investigators will conduct a three-arm mixed-methods randomized controlled trial (RCT) among 186 Chinese Childhood Cancer Survivors (CCCs). The three groups are VR hypnosis, cognitive behavioral therapy for insomnia (CBT-I), and VR relaxation. The VR hypnosis intervention contains six 30-minute sessions conducted by a clinical psychologist on 6 consecutive Saturdays in Hong Kong Children's Hospital (HKCH) or participants' home depend on participants' preference. Instead of treatment-as-usual and sleep hygiene groups, investigators will use the CBT-I as the active control because it is recommended as a first-line treatment for poor sleep. CBT-I group will have six 30-minute sessions in HKCH or home depend on participants' preference on six consecutive Saturdays. The VR relaxation group will allow us to distinguish the effects of VR from those of VR hypnosis, which has the same length and delivery mode as VR hypnosis, but without a hypnosis component. The study will be conducted at HKCH, which is the only hospital in HK that provides medical follow-ups for children with cancer. Data collection will be done at baseline, as well as immediately and 1, 3, and 6 months after completion of the intervention. Multiple assessment timepoints will capture changes over time.

ELIGIBILITY:
Inclusion Criteria:

* completed active cancer treatment for ≥1 month
* able to speak Cantonese and read Chinese
* aged 12-18 years
* poor sleeper as indicated by a PSQI score ≥ 5

Exclusion Criteria:

* Survivors with learning and/or behavioral problems in medical records and those who are using sleep medication and/or previously experienced any adverse events (e.g., headache and motion sickness) when using VR

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
subjective sleep quality | Baseline, immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  The 19-item Pittsburgh Sleep Quality Index (PSQI) will be used to assess participants' subjective sleep quality in the past month. Total scores range from 0 to 57. Poor sleepers have scores ≥ 5. The PSQI is reliable and valid to assess subjective sleep quality.

SECONDARY OUTCOMES:
total sleep time | Over a course of 7 days before the intervention begins, immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  All participants will wear the Actigraph wGT3X-BT to collect data on total sleep time.
sleep-onset latency | Over a course of 7 days before the intervention begins, immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  All participants will wear the Actigraph wGT3X-BT to collect data on sleep-onset latency.
sleep efficiency | Over a course of 7 days before the intervention begins, immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  All participants will wear the Actigraph wGT3X-BT to collect data on sleep efficiency.
awakening frequency after sleep onset | Over a course of 7 days before the intervention begins, immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  All participants will wear the Actigraph wGT3X-BT to collect data on awakening frequency after sleep onset.
sleep fragmentation index | Over a course of 7 days before the intervention begins, immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  All participants will wear the Actigraph wGT3X-BT to collect data on sleep fragmentation index.
brain electrophysiological activities | Two consecutive nights at baseline, during the intervention period (5 minutes before, during, and 5 minutes after hypnosis), one night immediately after completing the intervention, and one night at 6-month follow-up
  Participants in the VR hypnosis group will wear the Somté PSG under the supervision of a sleep technician. In the 6 hypnosis sessions, the electrophysiological record by the Somté PSG will occur. It aims to examine the changes in brain activities associated with hypnosis and explore how the changes may relate to alterations in brain electrophysiological activities in sleep. To record brain activities in sleep, participants in the VR hypnosis group will wear the Somté PSG at different time points.
usefulness | 6 months after completion of the intervention
  Participants in the VR hypnosis group will complete a validated questionnaire to assess perceived usefulness (6 items) of VR hypnosis. Higher scores reflect higher perceived usefulness which can reflect the technological challenges and predict the actual use of technology.
incremental cost-effectiveness ratio (ICER) | Immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  The cost-effectiveness of VR hypnosis is based on the cost divided by subject sleep quality gained and that divided by Quality-Adjusted Life Year (QALY) gained (derived from QoL).
depressive symptoms | Baseline, immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  The Center for Epidemiological Studies Depression Scale for Children (CES-DC) contains 20 items will be used to assess depressive symptoms. Total scores range from 0 to 60. Higher scores indicate more depressive symptoms. The psychometric properties of the CES-DC have been established in Chinese children with cancer.
cancer-related fatigue | Baseline, immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  The 12-item Fatigue Scale-Adolescent (FS-A) will be used to measure participants' cancer-related fatigue levels. Higher scores represent higher levels of fatigue. The FS-A is a reliable and valid measure for Chinese CCSs.
pain level | Baseline, immediately after completing the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  A visual analogue scale will be used to assess participants' pain levels. Participants will indicate their pain scores on a 100-mm horizontal line, with one end indicating no pain and another indicating the worst possible pain. This is a reliable and valid method for assessing pain in CCSs.
quality of life (QoL) | Baseline, on completion of the intervention, 1 month after completion of the intervention, 3 months after completion of the intervention, 6 months after completion of the intervention
  QoL will be assessed EuroQol five dimensions-youth version-3 level (EQ-5D-Y-3L). It contains five items evaluated on 3 levels. The score will be converted into a single utility score using a published algorithm. This scale was validated in Hong Kong Chinese adolescents, with the normative dataset being built.
ease of use | 6 months after completion of the intervention
  Participants in the VR hypnosis group will complete a validated questionnaire to assess perceived ease of use (6 items) of VR hypnosis. Higher scores reflect higher perceived ease of use which can reflect the technological challenges and predict the actual use of technology.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong